CLINICAL TRIAL: NCT04439786
Title: Efficacy of Intravenous Infusion of Lidocaine in Sedation for Colonoscopy: a Randomised Placebo-controlled Study
Brief Title: Intravenous Infusion of Lidocaine in Colonoscopy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, Vice president of Qilu Hospital, Shandong University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 2020SDU-QILU-021
Record Dates: First submitted 2020-06-18; First posted 2020-06-19 (Actual); Last update posted 2020-06-19 (Actual); Status verified 2020-06

CONDITIONS: Sedation
Keywords: intravenous lidocaine coloscopy
MeSH Terms: interventions — Sodium Chloride; Lidocaine

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to controll group or lidocaine group. Participants of control group are given placebo while participants of lidocaine group are given lidocaine.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Placebo Comparator): the control group will be given the same volume of saline as the experimental group
  Interventions: Drug: placebo
- lidocaine group (Experimental): the experimental group will be given l-1.5mg lidocaine and then 2mg/kg/h
  Interventions: Drug: lidocaine

INTERVENTIONS:
Drug: placebo — the control group will be given the same volume of saline.
  Other Names: saline
  Arms: control group
Drug: lidocaine — the experimental group will be given 1-1.5mg/kg lidocaine and then 2mg/kg/h
  Other Names: Compound Lidocaine Hydrochloride Injiection
  Arms: lidocaine group

SUMMARY:
intravenous infusion of lidocaine significantly reduce fatigue and pain and improve the patients satisfaction after sedation for colonoscopy.

DETAILED DESCRIPTION:
This study divide patients into two groups, lidocaine group one will be given lidocaine intravenously; control group will be given saline . the difference between patients fatigue and pain will be compared. and the propofol consumption, pain after infusion of propofol, patients, endoscopists and anaesthesist satifaction, the incidence of hypotenstion, hypoxia, and bradycardia will aslo be compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria: patients aged >18 years who were scheduled for colonscopy at Qilu hospital.

Exclusion Criteria:patients with ASA (American Society of Anesthesiologists) Class 4 or 5, pre-existing hypoxemia (SpO2 <90%), hypotension (systolic blood pressure <90 mm Hg), bradycardia (HR<50 beats/min), uncontrolled hypertension (SBP >170 mm Hg, diastolic blood pressure>100 mm Hg), severe renal or liver failure, pregnancy or lactation, allergy to lidocaine, atrioventricular block, epilepsy, and inability to give informed consen

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
fatigue score after colonoscopy | half a year
  fatigue were measured on a 0-10VAS at arrival in the recovery room ,30min later

SECONDARY OUTCOMES:
pain socre after colonoscopy | half a year
  pain were measured on a 0-10VAS at arrival in the recovery room ,30min later

OTHER OUTCOMES:
infusion pain when adminstrate propofol | half a year
  infusion pain was divided into no pain, mide pain and severe pain
Safety assessed by the rate of hypoxia during the procedure Safety assessed by the rate of hypoxia during the procedure | half a year
  Hypoxia, defined as peripheral oxygen saturation <90% for >10 seconds
Safety assessed by the rate of hypotention during the procedure | half a year
  Hypotension, defined as systolic blood pressure <90 mmHg
Safety assessed by the rate of breadycardia during the procedure | half a year
  Bradycardia, defined as heart rate <50 beats/min
Safety assessed by the rate of required airway management during the procedure | half a year
  Required airway management such as jaw lifting, mask ventilation, or tracheal intubation in severe hypoxia Required airway management such as jaw lifting, mask ventilation, or tracheal intubation in severe hypoxia
Safety assessed by the rate of involuntary movement | half a year
  Involuntary movements, defined as unconscious movements requiring restraint or severe limb movement
endoscopists satisfaction assessed by the performer | half a year
  the endoscopists satisfacition score were assessed on a 0-10VAS after the procedure
patient satisfaction assessed by the patient | half a year
  the patient satisfacition score were assessed on a 0-10VAS 30mins after the procedure
anesthetist satisfaction assessed by the anesthestist | half a year
  the anesthetist satisfacition score were assessed on a 0-10VAS after the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Shan dong China, Study Chair — Qilu Hospital of Shandong University
Locations (1):
- Department of Gastroenterology, Qilu Hospital, Shandong University, Jinan, Shandong, China